CLINICAL TRIAL: NCT02015520
Title: A Phase IIb, Randomized, Multi-Center, Double-Blind, Dose-Ranging Study to Evaluate the Efficacy and Safety of Clazakizumab in Subjects With Moderate to Severe Active Rheumatoid Arthritis Who Have Experienced an Inadequate Response to TNF Inhibitors
Brief Title: Phase IIB Dose Ranging Study in Subjects With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM133-066; 2013-003780-65 (EudraCT Number)
Record Dates: First submitted 2013-12-06; First posted 2013-12-19 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Clazakizumab (Dose # A) (Double-Blind) (Experimental): Clazakizumab Dose # A injection by subcutaneous for 12 weeks + background Methotrexate
  Interventions: Drug: Clazakizumab
- Arm 2: Clazakizumab (Dose # B) (Double-Blind) (Experimental): Clazakizumab Dose # B injection by subcutaneous for 12 weeks + background Methotrexate
  Interventions: Drug: Clazakizumab
- Arm 3: Clazakizumab (Dose # C) (Double-Blind) (Experimental): Clazakizumab Dose # C injection by subcutaneous for 12 weeks + background Methotrexate
  Interventions: Drug: Clazakizumab
- Arm 4: Placebo matching with Clazakizumab (Double-Blind) (Experimental): Clazakizumab Dose # D injection by subcutaneous for 12 weeks + background Methotrexate
  Interventions: Drug: Placebo (Matching with Clazakizumab)

INTERVENTIONS:
Drug: Clazakizumab
  Other Names: BMS-945429
  Arms: Arm 1: Clazakizumab (Dose # A) (Double-Blind); Arm 2: Clazakizumab (Dose # B) (Double-Blind); Arm 3: Clazakizumab (Dose # C) (Double-Blind)
Drug: Placebo (Matching with Clazakizumab)
  Arms: Arm 4: Placebo matching with Clazakizumab (Double-Blind)

SUMMARY:
The primary purpose of this study is to identify an appropriate dose of study medication.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Diagnosis of active Rheumatoid Arthritis (RA) by standard criteria (American Rheumatism association (ARA) [1987] or American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) [2010]) at least 16 weeks prior to screening
* ACR global functional status class of 1 to 3
* Documented evidence of inadequate response tumor necrosis factor (TNF) inhibitors
* All subjects must have been receiving treatment with a minimum dose of 15 mg per week of Methotrexate for at least 12 weeks and at a stable dose for 28 days prior to screening. A dose as low as 10 mg Methotrexate is permitted if 15 mg could not be reached, due to toxicity. In Japan, Korea and Taiwan, a minimum dose of 7.5 mg per week is permitted. Additional treatment with Hydroxychloroquine or Chloroquine is permitted, if it is at a dose approved for the treatment of RA and the dose has been stable for at least 28 days prior to screening
* Minimum of 6 swollen and 6 tender joints on a 66/68 joint count at screening and at baseline (Day 1)
* Elevated High-sensitivity (hs) CRP and/or ESR

Exclusion Criteria:

* Active serious infection
* History of or active tuberculosis (TB)
* Elevated liver function tests (LFTs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (21):
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - Mercy Clinic Hot Springs Communities, Hot Springs, Arkansas
  - Valerius Med Group & Res Ctr Of Greater Long Beach, Inc., Long Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Joint And Muscle Medical Care And Research Institute (Jmmcri), Charlotte, North Carolina
  - Physicians East, Pa, Greenville, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Arthritis & Rheumatology Center Of Oklahoma Pllc, Oklahoma City, Oklahoma
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Low Country Rheumatology, Charleston, South Carolina
  - Rheumatology Consultants Pllc, Knoxville, Tennessee
  - Center For Inflammatory Disease, Nashville, Tennessee
  - Seattle Rheumatology Associates, Seattle, Washington
- Argentina (4):
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Buenos Aires
  - Local Institution, Córdoba
  - Local Institution, San Miguel de Tucumán
- Canada (3):
  - Cividino Medicine Professional Corporation, Hamilton, Ontario
  - Credit Valley Rheumatology, Mississauga, Ontario
  - Dr. Latha Naik Medical Professional Corporation, Saskatoon, Saskatchewan
- France (3):
  - Local Institution, Bordeaux
  - Local Institution, Paris
  - Local Institution, Poitiers
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Veszprém
- Italy (4):
  - Local Institution, Catanzaro
  - Local Institution, Florence
  - Local Institution, Napoli
  - Local Institution, Pisa
- Japan (8):
  - Local Institution, Chiba, Chiba
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Kato-shi, Hyōgo
  - Local Institution, Nagano, Nagano
  - Local Institution, Sasebo-shi, Nagasaki
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Toshima-ku, Tokyo
  - Local Institution, Nishimura, Wakayama
- Mexico (5):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Mérida, Yucatán
  - Local Institution, Guadalajara
  - Local Institution, San Luis Potosí City
- South Africa (2):
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Stellenbosch, Western Cape

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Methotrexate (MTX): Placebo (5% dextrose) subcutaneous (SC) administration once every 4 weeks for 12 weeks plus background methotrexate (MTX)
- Clazakizumab (1 mg) + MTX: Clazakizumab (1 mg) SC administration once every 4 weeks for 12 weeks + background Methotrexate
- Clazakizumab (5 mg) + MTX: Clazakizumab (5 mg) SC administration once every 4 weeks for 12 weeks + background Methotrexate
- Clazakizumab (25 mg) + MTX: Clazakizumab (25 mg) SC administration once every 4 weeks for 12 weeks + background Methotrexate
Period: Overall Study
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Started | 40 | 21 | 42 | 40
Completed | 35 | 17 | 35 | 36
Not Completed | 5 | 4 | 7 | 4
Not completed — Lack of Efficacy | 1 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Subject Request to Discontinue Study Treatment | 1 | 1 | 2 | 1
Not completed — Subject no Longer Meets Study Criteria | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX | Total
Number analyzed (Participants) | 40 | 21 | 42 | 40 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 15 | 35 | 32 | 114
  >=65 years | 8 | 6 | 7 | 8 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.21) | 55.8 (11.20) | 53.4 (13.75) | 52.6 (13.21) | 53.8 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 18 | 33 | 35 | 121
  Male | 5 | 3 | 9 | 5 | 22
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 3 | 0 | 5
  Argentina | 4 | 4 | 4 | 6 | 18
  Hungary | 7 | 3 | 7 | 5 | 22
  United States | 11 | 7 | 11 | 9 | 38
  Japan | 4 | 3 | 5 | 4 | 16
  Italy | 1 | 0 | 0 | 0 | 1
  Mexico | 8 | 1 | 8 | 12 | 29
  South Africa | 4 | 2 | 2 | 4 | 12
  France | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score in 28 Joints - C-reactive Protein (DAS28-CRP) at Week 12
Description: DAS28-CRP describes severity of rheumatoid arthritis. The components of the joint count assessment are shoulder, elbow, wrist, metacarpophalangeal joints 1 through 5, proximal interphalangeal joints 1 through 5, and the knee joints on the right and left sides, whereby the number of affected joints, tender and swollen, respectively, are counted. The formula used to calculate the score is: DAS28-CRP=0.56 \times \sqrt{TEN28} + 0.28 \times \sqrt{SW28} + 0.36 \times \ln(CRP+1) + 0.014 \times SA+0.96 with:
  TEN28: number of joints with tenderness upon touching SW28: number of swollen joints CRP: C-reactive Protein SA: subjective assessment of disease activity by the patient during the preceding 7 days on a scale between 0 and 100 ("0":no activity, "100": highest activity possible).
  DAS-CRP score range is 0.49 to 9.07 A DAS-CRP value >5.1 corresponds to a high disease activity A DAS-28 reduction by 0.6 represents a moderate improvement. A reduction >1.2 represents a major improvement
Time Frame: Baseline and Week 12
Population: Modified Intent-to-Treat (mITT) Analysis Population: All randomized subjects who received at least 1 dose of the study medication.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 34 | 15 | 35 | 37
score on a scale | -0.75 (0.22) | -1.10 (0.33) | -2.10 (0.22) | -2.43 (0.22)
Statistical Analysis 1: Comparison: Placebo + Methotrexate (MTX) vs Clazakizumab (1 mg) + MTX; Test type: Superiority; p = 0.38, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo + Methotrexate (MTX) vs Clazakizumab (5 mg) + MTX; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo + Methotrexate (MTX) vs Clazakizumab (25 mg) + MTX; Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: American College of Rheumatology (ACR) 20/50/70 Response Rates
Description: The ACR20/50/70 is a composite measure defined as both improvement of 20%, 50% or 70% in the number of tender and number of swollen joints, and a 20%, 50% or 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Time Frame: At week 12
Population: mITT
Measure: Number; unit: percentage of responders
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 40 | 21 | 42 | 40
percentage of responders
  ARC20 responders | 27.5 | 14.3 | 50.0 | 47.5
  ARC50 responders | 7.5 | 14.3 | 21.4 | 22.5
  ARC70 responders | 2.5 | 4.8 | 9.5 | 15.0

3. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Week 12
Description: CDAI is a composite index for assessing disease activity. CDAI is based on the simple summation of the count of swollen joint count (SCJ) (0-28) and tender joint count (TJC) (0-28) along with patient global assessment (0-10) Scale and physician global assessment (0-10) for estimating disease activity where 10 means maximal activity. The CDAI has a range from 0 to 76.
  CDAI <= 2.8 = Remission CDAI > 2.8 and <= 10 = Low Disease Activity CDAI > 10 and <= 22 = Moderate Disease Activity CDAI > 22 = High Disease Activity
Time Frame: Baseline and week 12
Population: mITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 32 | 14 | 36 | 37
score on a scale | -9.9 (2.656) | -12.8 (3.961) | -17.4 (2.545) | -21.6 (2.539)

4. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Week 12
Description: SDAI is a composite index for assessing disease activity. CDAI is based on the simple summation of the count of swollen joint count (0-28) and tender joint count (0-28) along with patient global assessment (0-10) Scale and physician global assessment (0-10) for estimating disease activity where 10 means maximal activity and C-reactive protein (0-10). The SDAI has a range from 0 to 86.
  0.0 - 3.3 = Remission 3.4 - 11.0 = Low Activity 11.1 - 26.0 = Moderate Activity 26.1 - 86.0 = High Activity
Time Frame: Baseline and week 12
Population: mITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 32 | 14 | 35 | 37
score on a scale | -9.68 (2.6846) | -13.08 (4.0011) | -20.15 (2.5928) | -24.02 (2.5677)

5. Secondary Outcome: Boolean Remission at Week 12
Description: Boolean-based definition:
  At any time point, a patient must satisfy all of the following:
  TJC ≤1 (0-28) SJC ≤1 (0-28) CRP ≤1 mg/dl Patient Global Assessment ≤1 (on a 0-10 scale)
Time Frame: At week 12
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 40 | 21 | 42 | 40
percentage of participants | 5.0 | 4.8 | 2.4 | 5.0

6. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 12
Description: Patients report the amount of difficulty they have in performing 8 categories. Each category is scored on a scale ranging from 0 (performed without any difficulty) to 3 (cannot be done at all). The HAQ-DI is then calculated by summing the scores and dividing by the number of categories answered. Total score is between 0-3.0. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment. The HAQ-DI cannot be calculated if the subject does not have scores for at least 6 categories. A response was defined as a subject with a reduction from baseline in HAQ-DI of at least 0.22.
Time Frame: Baseline and Week 12
Population: mITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 35 | 16 | 36 | 36
score on a scale | -0.25 (0.0906) | -0.09 (0.1307) | -0.31 (0.0889) | -0.46 (0.0905)

7. Secondary Outcome: Percent of Participants With a DAS28-Erythrocyte Sedimentation Rate (ESR) <2.6
Description: DAS28- ESR = Disease Activity Scores 28 based on erythrocyte sedimentation rate. A DAS28-ESR below 2.6 is interpreted as remission.
Time Frame: At week 12
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 40 | 21 | 42 | 40
percentage of participants | 2.5 | 4.8 | 7.1 | 15.0

8. Secondary Outcome: Percent of Participants With a DAS28-C Reactive Protein (CRP) <2.6
Description: DAS28-CRP = Disease Activity Scores 28 based on C Reactive Protein. A DAS28-CRP below 2.6 is interpreted as remission.
Time Frame: At week 12
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
Number analyzed (Participants) | 40 | 21 | 42 | 40
percentage of participants | 5.0 | 9.5 | 14.3 | 15.0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks for each participant
Description: As-Treated Analysis Population: All subjects who received at least 1 dose of study medication.
Arm/Group | Placebo + Methotrexate (MTX) | Clazakizumab (1 mg) + MTX | Clazakizumab (5 mg) + MTX | Clazakizumab (25 mg) + MTX
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/21 | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/21 | 0/42 | 1/40
Other Adverse Events (participants affected / at risk) | 14/40 | 5/21 | 24/42 | 28/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Methotrexate (MTX) (N=40) | Clazakizumab (1 mg) + MTX (N=21) | Clazakizumab (5 mg) + MTX (N=42) | Clazakizumab (25 mg) + MTX (N=40)
SUDDEN DEATH (General disorders) | 1 | 0 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Methotrexate (MTX) (N=40) | Clazakizumab (1 mg) + MTX (N=21) | Clazakizumab (5 mg) + MTX (N=42) | Clazakizumab (25 mg) + MTX (N=40)
NASOPHARYNGITIS (Infections and infestations) | 3 | 0 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 2 | 1
BRONCHITIS (Infections and infestations) | 0 | 1 | 1 | 1
SINUSITIS (Infections and infestations) | 2 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1 | 1
FATIGUE (General disorders) | 1 | 1 | 2 | 0
INJECTION SITE REACTION (General disorders) | 0 | 0 | 1 | 3
INJECTION SITE RASH (General disorders) | 1 | 1 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 2 | 0
CONTUSION (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 2
DIZZINESS (Nervous system disorders) | 2 | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 2 | 0
ORAL HERPES (Infections and infestations) | 2 | 0 | 0 | 0
EAR INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 1
LABYRINTHITIS (Infections and infestations) | 0 | 0 | 0 | 1
SKIN CANDIDA (Infections and infestations) | 0 | 0 | 0 | 1
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 0 | 1 | 1
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1 | 1
BLOOD UREA INCREASED (Investigations) | 0 | 0 | 1 | 0
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 0 | 0 | 1 | 0
NEUTROPHIL COUNT INCREASED (Investigations) | 1 | 0 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 1 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 1 | 0
TENSION HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1
TREMOR (Nervous system disorders) | 0 | 0 | 1 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 0 | 2 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0
SECONDARY HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 0
EYE PAIN (Eye disorders) | 0 | 0 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 1 | 0
VULVOVAGINAL DISCOMFORT (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
AXILLARY PAIN (General disorders) | 0 | 0 | 1 | 0
DRUG INTOLERANCE (General disorders) | 1 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 0 | 0
INJECTION SITE BRUISING (General disorders) | 0 | 1 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 1
INJECTION SITE PRURITUS (General disorders) | 0 | 0 | 0 | 1
INJECTION SITE VESICLES (General disorders) | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 1 | 0
VACCINATION SITE REACTION (General disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No